CLINICAL TRIAL: NCT00165685
Title: A Double-Blind, Placebo-Controlled, Comparative Study of KES524 in Patients With Obesity Disease
Brief Title: A Comparative Study of KES524 in Patients With Obesity Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KES524-J081-161
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

INTERVENTIONS:
Drug: Sibutramine Hydrochloride Monohydrate

SUMMARY:
To investigate the efficacy and safety of KES524 in patients with obesity (visceral fat obesity with type 2 diabetes and dyslipidemia), a 52-week, double-blind, placebo-controlled comparative study is conducted. This study aims to examine superiority of KES524 to placebo by employing change and percent change in body weight (primary endpoints) and changes in proportion of subjects achieving ≧ 5% weight reduction, BMI, waist circumference, visceral fat area, subcutaneous fat area, V/S ratio by abdominal CT scan, HbA1c, TG and HDL-C (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≧25 kg/m2 of BMI at the start of the observation period
* Patients with visceral fat area ≧100 cm2 measured with abdominal CT scan
* Patients with the following two health impairments:

  1. Patients with previously diagnosed type 2 diabetes and HbA1c between ≧6.1% and <9.0% at the start of observation period
  2. Patients with ≧150 mg/dL of triglyceride (TG), and/or <40 mg/dL of high-density lipoprotein cholesterol (HDL-C) for serum lipid parameters as dyslipidemic index at the start of the observation period
* Patients continuously receiving diet therapy for 8 weeks or longer before the start of the observation period
* Patients not receiving antidiabetic (12 weeks), antihyperlipidemics (4 weeks) and/or antihypertensive (4 weeks) drugs. If used, those who have received a consistent dosage and administration beginning more than 4 weeks (more than 12 weeks for antidiabetics) before the start of the observation period
* Patients with ambulatory treatment aged between ≧20 years and <65 years at the time of obtaining informed consent
* Patients who are given full explanation about the study objective and contents and can give written informed consent

Exclusion Criteria:

* Patients with pulse rate of ≧100/min during the observation period
* Patients with systolic blood pressure of ≧160 mmHg and/or with diastolic blood pressure of ≧100 mmHg during the observation period
* Patients with body weight loss of ≧3% as compared to that at the start of the observation period, or body mass index (BMI) that is reduced to <25 kg/m2 during the observation period
* Patients who have received insulin within 12 weeks before the start of the observation period
* Patients with present illness or past history of severe eating disorder (e.g., anorexia nervosa or bulimia nervosa)
* Patients with present illness or past history of drug allergy or severe allergic disease(s)
* Patients with present illness or past history of the following disorders:
* Coronary artery disease (myocardial infarction, angina), heart failure
* Serious diseases such as cardiovascular (severe tachycardiac heart failure), renal (renal failure), hepatic (severe hepatitis, cirrhosis), pancreatic (severe pancreatitis), psychotic (severe depression, schizophrenia, alcohol addict, drug addict) disorders
* Pregnant or lactating women, or women who intend to become pregnant during the study period
* Patients who previously participated in and were treated in another clinical study of KES524
* Patients who have received another study drug within 24 weeks before starting observation period of this study
* Patients who are judged to be ineligible for study entry by the investigator or subinvestigator

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change and percent change in body weight

SECONDARY OUTCOMES:
Proportion of subjects achieving ≧5% weight reduction
Change in BMI
Change in waist circumference
Change in visceral fat area, subcutaneous fat area, and V/S ratio by abdominal CT scan
Change in HbA1c
Change and percent change in fasting serum lipids (TG, HDL-C)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Takeuchi, Study Director — Development Clinical Research Dept., Clinical Research Center
Locations (18):
- Japan (18):
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Fukushima, Fukushima
  - Kōriyama, Fukushima
  - Maebashi, Gunma
  - Hitachiota, Ibaraki
  - Mito, Ibaraki
  - Naka, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Sendai, Miyagi
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Hachiōji, Tokyo
  - Itabashi-ku, Tokyo
  - Minato-ku, Tokyo
  - Shibuya-ku, Tokyo